CLINICAL TRIAL: NCT06456619
Title: Clinical and Radiographic Evaluation of Composite Resin Restorations and Computer-Aided Restorations in Young Permanent Molar Teeth With Molar Incisor Hypomineralization
Brief Title: CAD-CAM or Adhesive Approaches for MIH Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-KA19/04
Record Dates: First submitted 2024-05-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Molar Hypomineralization; Dental Restoration Failure of Marginal Integrity
Keywords: Molar incisor hypomineralization; CAD-CAM supported restoration; Composite resin restoration
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: Observational clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Composite resin (Filtek Z250, 3M ESPE) (Active Comparator): A pretreatment protocol including sodium hypochlorite and ortho-phosphoric acid was applied to the tooth surface. Then, the tooth was restored with a composite resin material (Filtek Z250, 3M ESPE). This protocol is a clinically approved way for restoring hypomineralized teeth.
  Interventions: Other: Tooth restoration
- CAD-CAM supported (Cerasmart, GC Dental) (Experimental): The preparation was completed by making bevels on the enamel surfaces. Then, an intraoral impression was taken to sent to the laboratory for manufacturing CAD-CAM-supported restoration with a nanohybrid ceramic material (Cerasmart, GC Dental). CAD-CAM supported restorations can be done by using a lot of restorative blocks by milling them. In this study, we preferred using resin-based blocks (Cerasmart, GC Dental) to compare with the control group.
  Interventions: Other: Tooth restoration

INTERVENTIONS:
Other: Tooth restoration — Comparison of composite resin and CAD-CAM supported restorations for hypomineralized molar teeth in children

SUMMARY:
Aim: This randomized controlled clinical study aimed to compare direct composite resin restorations and Computer Aided Design-Computer Aided Manufacturing (CAD-CAM) supported inlay or onlay restorations in young permanent molar teeth with hypomineralization.

The main questions aim to answer are:

* The clinical success rate of CAD-CAM supported restorations
* The highest clinical success rate for restoring hypomineralized teeth.

Materials and method: Children aged 6-14 years old without any systemic conditions with 32 first and second hypomineralized permanent molar teeth were included in the study. Patients were randomly distributed into 2 groups as direct composite resin restorations and CAD-CAM supported inlay or onlay restorations. All restored teeth were evaluated clinically and radiographically for 24-months. Statistical significance was accepted as p<0.05.

DETAILED DESCRIPTION:
After randomization and local anesthesia administration, caries removal and preparation were completed under rubber-dam isolation. After preparation, 60 seconds of orthophosphoric acid, 60 seconds of 5% sodium hypochlorite and 30 seconds of orthophosphoric acid steps were applied before bonding agent and composite resin restorations. On the other hand, the preparation was completed by making a bevel on the enamel surfaces and a nanohybrid ceramic material used for the manufacturing CAD-CAM supported inlay or onlay restorations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first and second permanent molar teeth that have loss of more than one surface due to hypomineralization and seen with white, brown, or yellow opacities on anterior permanent teeth
* Patients without any systemic, physical, physiological, or allergic conditions

Exclusion Criteria:

* Patients who had symptoms during the follow-up periods
* Patients who did not attend follow-up appointments

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation (Modified USPHS criteria- Anatomic form) | 24 months
  Anatomic form was examined by inspection at 3,6,12,18, and 24 months.
Clinical evaluation (Modified USPHS criteria-Surface roughness) | 24 months
  Surface roughness was examined by inspection and probing at 3,6,12,18, and 24 months.
Clinical evaluation (Modified USPHS criteria-Marginal adaptation) | 24 months
  Marginal adaptation was examined by inspection and probing at 3,6,12,18, and 24 months.
Clinical evaluation (Modified USPHS criteria-Marginal discoloration) | 24 months
  Marginal discoloration was examined by inspection at 3,6,12,18, and 24 months.
Clinical evaluation (Modified USPHS criteria-Retention) | 24 months
  Retention was examined by inspection and probing at 3,6,12,18, and 24 months.
Clinical evaluation (Modified USPHS criteria-Color stability) | 24 months
  Color stability was examined by inspection at 3,6,12,18, and 24 months.
Clinical evaluation (Modified USPHS criteria-Secondary caries) | 24 months
  Secondary caries was examined by inspection and probing at 3,6,12,18, and 24 months.
Clinical evaluation (Modified USPHS criteria-Proximal contact) | 24 months
  Proximal contact was examined by inspection and probing at 3,6,12,18, and 24 months.
Radiographical evaluation (Lamina dura) | 24 months
  Lamina dura continuity was evaluated by periapical radiographs taken at 6, 12, 18, and 24-months.
Radiographical evaluation (Change in inter-root trabeculation continuity) | 24 months
  Change in inter-root trabeculation continuity was evaluated by periapical radiographs taken at 6, 12, 18, and 24-months.
Radiographical evaluation (Radiolucent area development) | 24 months
  Radiolucent area development in the inter-root area was evaluated by periapical radiographs taken at 6, 12, 18, and 24-months.

CONTACTS AND LOCATIONS:
Overall Officials: Didem Sakaryalı Uyar, PhD MD, DDS, Principal Investigator — Başkent Universiry
Locations (1):
- Başkent University, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Information about patients might be requested from the principal author due to reasonable cause.